CLINICAL TRIAL: NCT04987684
Title: Objective Measures of Cochlear Implant Electrode Position and Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sophie McKenny (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor-Investigator, Sophie McKenny, Clinical Researcher, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 285894
Record Dates: First submitted 2020-09-25; First posted 2021-08-03 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Cochlear Implants
Keywords: cochlear implant; electrophysiology; auditory nerve fibres; extra cochlear electrodes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of Care (Other)
  Interventions: Diagnostic Test: SCINSEV and PECAP

INTERVENTIONS:
Diagnostic Test: SCINSEV and PECAP — To measure PECAP and SCINSEVs. To find whether electrodes are outside of the cochlear or within dead regions within the cochlear.

SUMMARY:
Recruit adult patients eligible for cochlear Implant surgery. During routine surgery monitor electrode placement with new 'SCINSEV' technique and complete 'PECAPs' on patient to identify if any of the electrodes have misplaced.

Follow up with patient after surgery for post operative appointment with same measurements.

DETAILED DESCRIPTION:
Cochlear implants (CIs) restore hearing to deaf patients by electrically stimulating the auditory nerve using an array of electrodes inserted into the cochlea (inner ear). All electrodes should be successfully inserted in the cochlea, with each electrode exciting a discrete range of auditory nerve fibers.

Our research investigates two exceptions to this ideal situation, both of which impair the participant's ability to clearly hear sounds such as speech. One exception occurs when some electrodes are located outside the cochlea, limiting the amount of information that is conveyed to the brain and potentially causing unwanted side effects.

Our research will identify these extra-cochlear electrodes during the CI operation, by stimulating each electrode in turn and recording from all other electrodes.

This "SCINSEV" technique then uses a sophisticated computational method to identify which if any electrodes are out of the cochlea. Even when all electrodes are in the cochlea, however, some may produce broad current spreads, which will "blur" the perception of sounds. Our second "PECAP" method measures these instances by stimulating pairs of electrodes and recording the neural responses. It also uses a new computational method, this time so as to calculate the neural spread from each electrode.

Both methods use fast, non-invasive, objective measurements that use the built-in capabilities of the implant .The interventions used are very similar to those employed in standard clinical practice, and the results will pave the way for better identification and management of poor hearing by CI patients

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing or able to consent to participation in the study
* Meets normal candidacy requirements for cochlear implantation
* At least 18 years of age at time of consent being given
* Patent cochlea as verified by CT or MRI scan
* No additional complex needs that would prevent study procedures being followed
* Agreement to participate in the study

Exclusion Criteria:

* Using medication in a manner that might affect hearing levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Validation of extra cochlear electrodes | 12 months
  Number of extra-cochlear electrodes obtained using our "SCINSEV" analysis correspond to the actual number of extra-cochlear electrodes observed during different stages of insertion.

SECONDARY OUTCOMES:
Pre and post op loudness comparison | 12 months
  Numbers of neural dead regions and wide current spread estimated intra-operatively and using equal current per electrode using our "PECAP" method correspond to those occurring post-operatively and using equal loudness per electrode

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Borsetto, Principal Investigator — Addenbrookes Hospital, CUH
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided